CLINICAL TRIAL: NCT00879359
Title: A Phase II Trial of a Vascular Endothelial Growth Factor (VEGF) Monoclonal Antibody, AVASTIN, in Combination With Cytotoxic Chemotherapy CARBOPLATIN and PACLITAXEL for Recurrent/Advanced Endometrial Cancer
Brief Title: Trial of Vascular Endothelial Growth Factor (VEGF), Bevacizumab, in Combination With Cytotoxic Chemotherapy for Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20806
Record Dates: First submitted 2009-04-09; First posted 2009-04-10 (Estimated); Results first posted 2017-04-26 (Actual); Last update posted 2017-04-26 (Actual); Status verified 2017-03

CONDITIONS: Endometrial Carcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Carboplatin; Paclitaxel; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- I (Experimental)
  Interventions: Drug: carboplatin, paclitaxel, and bevacizumab

INTERVENTIONS:
Drug: carboplatin, paclitaxel, and bevacizumab — All patients enrolled will receive carboplatin AUC 5 plus paclitaxel 175 mg/m2 (135 mg/m2 if prior radiation to greater than 25% of bone marrow) plus bevacizumab 15 mg/kg every 3 weeks.
  Other Names: Avastin

SUMMARY:
The purpose of this study is to find out whether the addition of a drug called Avastin (avastin) to the two-drug combination of carboplatin and paclitaxel shrinks tumors better than the two-drug combination alone in the treatment of endometrial cancer. Avastin is a humanized monoclonal antibody (a type of protein that is normally made by the immune system to help defend the body from infection and cancer) produced by Genentech, Inc. Avastin is an antibody directed against vascular endothelial growth factor, or VEGF. VEGF is a potent, specific growth factor with a well defined role in normal and abnormal blood vessel formation. It is present in a wide variety of normal tissues, but is produced in excess by most solid cancers (tumors). In the setting of cancer, VEGF promotes the growth of blood vessels that feed the tumor cells.

DETAILED DESCRIPTION:
Exclusion Criteria

Disease-Specific Exclusions

* Patients with a concomitant malignancy other than non-melanoma skin cancer. Patients with a prior malignancy who have been disease-free for greater than 5 years or who received prior chemotherapy for that malignancy.
* Patients in whom pathological confirmation of the tumor is not obtainable. General Medical Exclusions
* Patients with concomitant medical illness such as serious uncontrolled infection, uncontrolled angina, or serious peripheral neuropathy, which, in the opinion of the treating physician, make the treatments prescribed on this study unreasonably hazardous for the patient.
* Patients with third degree or complete heart block are not eligible unless a pacemaker is in place. Patients on medications which alter cardiac conduction, such as digitalis, beta-blockers, or calcium channel blockers, or who have other conduction abnormalities or cardiac dysfunction may be placed on study at the discretion of the investigator.
* Patients whose circumstances will not permit study completion or adequate follow-up.
* Patients who are sensitive to E. Coli-derived drug preparations.
* Life expectancy of less than 12 weeks.
* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study other than a Genentech-sponsored avastin cancer study.
* Inadequately controlled hypertension (defined as systolic blood pressure greater than 150 and/or diastolic blood pressure greater than 100 mmHg on antihypertensive medications).
* Any prior history of hypertensive crisis or hypertensive encephalopathy.
* New York Heart Association (NYHA) Grade II or greater congestive heart failure (see Appendix C).
* History of myocardial infarction or unstable angina within 6 months prior to study enrollment.
* History of stroke or transient ischemic attack within 6 months prior to study enrollment.
* Known CNS disease.
* Significant vascular disease (e.g., aortic aneurysm, aortic dissection). Symptomatic peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy. Blood coagulation parameters: PT such that international normalized ratio (INR) is less than 1.5 (or an in range INR, between 2 and 3, if a patient is on a stable dose of therapeutic warfarin) and a PTT less than 1.5 times the institutional upper limit of normal.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study enrollment or anticipation of need for major surgical procedure during the course of the study.
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to study enrollment.

-History of abdominal fistula, gastrointestinal perforation, or intra- abdominal abscess within 6 months prior to study enrollment. Patients with clinical symptoms or signs of gastrointestinal obstruction and who require parenteral hydration and/or nutrition.

* Serious, non-healing wound, ulcer, or bone fracture.
* Proteinuria at screening as demonstrated by:
* Urine protein:creatinine (UPC) ratio greater than or equal to 1.0 at screening
* Known hypersensitivity to any component of avastin.
* Pregnant (positive pregnancy test) or lactating. Refusal to use of effective means of contraception (men and women) in subjects of child-bearing potential.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed primary Stage III or Stage IV (see FIGO staging-Appendix I) or recurrent endometrial carcinoma with MEASURABLE disease whose potential for cure by radiation therapy or surgery alone or in combination is very poor. Recurrent disease must be biopsy confirmed.
* Patients may have received prior cytotoxic chemotherapy

  (1 therapy) excluding a platinum/taxane. Patients may have received prior hormonal therapy or therapy with biologic agents, but such therapies must be discontinued 4 weeks prior to entry on this study.
* Patients in whom both radiation and chemotherapy is planned may receive radiation prior to entry on this study (order not specified). At least four weeks should have elapsed since completion of RT involving the whole pelvis or over 50% of the spine.
* Patients must be 18 years of age or older.

Exclusion Criteria:

* Patients with a concomitant malignancy other than Genentech, Inc Page 27 of 62 Bevacizumab Protocol 03-10-08 Page 27 non-melanoma skin cancer. Patients with a prior malignancy who have been disease-free for < 5 years or who received prior chemotherapy for that malignancy.
* Patients in whom pathological confirmation of the tumor is not obtainable.
* Patients with concomitant medical illness such as serious uncontrolled infection, uncontrolled angina, or serious peripheral neuropathy, which, in the opinion of the treating physician, make the treatments prescribed on this study unreasonably hazardous for the patient.
* Patients with third degree or complete heart block are not eligible unless a pacemaker is in place. Patients on medications which alter cardiac conduction, such as digitalis, beta-blockers, or calcium channel blockers, or who have other conduction abnormalities or cardiac dysfunction may be placed on study at the discretion of the investigator.
* Life expectancy of less than 12 weeks.
* Patients who are sensitive to E. Coli-derived drug preparations.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study enrollment or anticipation of need for major surgical procedure during the course of the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-12; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rose, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Maintenance Therapy With Bevacizumab: A phase II trial was conducted in patients with measurable disease. Paclitaxel (175 mg/m^2/3 hours), carboplatin (AUC 5) and bevacizumab (15 mg/kg) were administered q21 days. Patients in a complete response after 6 or 8 cycles received maintenance therapy with bevacizumab 15 mg/kg q21 days for 16 cycles.
Period: Overall Study
Arm/Group | Maintenance Therapy With Bevacizumab
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Maintenance Therapy With Bevacizumab
Number analyzed (Participants) | 15
Age, Continuous [Median (Full Range); unit: years] | 63 [32 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15
Stage (FIGO 2009) [Count of Participants; unit: Participants]
  IA | 4
  IB | 1
  IIB | 1
  IIIC1 | 1
  IIIC2 | 1
  IVB | 7
Tumor histology and grade [Count of Participants; unit: Participants]
  Serous papillary | 6
  Endometrioid grade 2 | 5
  Endometrioid grade 3 | 3
  Clear cell | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Progression Free Survival (PFS=Date of Progression of Disease or Death) at 6 Months Using Bevacizumab, Carboplatin, and Paclitaxel in Patients With Measurable Disease for Advanced/Recurrent Endometrial Cancer
Description: Number of patients with progression free survival measured at 6 months. Progression is defined using Response Evaluation Criteria in Solid Tumors Criteria (RECIST version 1.0), as a 20% increased in the sum of the longest diameter of target lesions, or a measure increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 58 months
Measure: Count of Participants; unit: Participants
Groups:
- Maintenance With Bevacizumab: carboplatin, paclitaxel, and bevacizumab: All patients enrolled will receive carboplatin AUC 5 plus paclitaxel 175 mg/m2 (135 mg/m2 if prior radiation to greater than 25% of bone marrow) plus bevacizumab 15 mg/kg every 3 weeks.
Arm/Group | Maintenance With Bevacizumab
Number analyzed (Participants) | 15
Participants
  Participants with PFS at 6 months | 14
  Partipants with progression at 6 months | 1
Statistical Analysis 1: Comparison: Maintenance With Bevacizumab; Test type: Superiority or Other; Hazard Ratio, log = 92, 95% CI 2-sided [64 to 99]

2. Secondary Outcome: Median Progression Free Survival of This Treatment Regimen in Patients With Advanced/Recurrent Endometrial Cancer.
Description: Median progression free survival measured in months. Progression of disease is defined using Response Evaluation Criteria in Solid Tumors Criteria (RECIST version 1.0), as a 20% increased in the sum of the longest diameter of the target lesions, or a measurable increased in a non-target lesion, or the appearance of a new lesion.
Time Frame: 58 months
Measure: Median (Full Range); unit: months
Groups:
- Maintenance Therapy With Bevacizumab: A phase II trial was conducted in patients with measurable disease. Paclitaxel (175 mg/m2/3 hours), carboplatin (AUC 5) and bevacizumab (15 mg/kg) were administered q21 days. Patients in a complete response after 6 or 8 cycles received maintenance therapy with bevacizumab 15 mg/kg q21 days for 16 cycles.
Arm/Group | Maintenance Therapy With Bevacizumab
Number analyzed (Participants) | 15
months | 18 [7 to 58]

3. Secondary Outcome: Number of Participants With Adverse Events Grades 1-5
Description: Toxicity and safety was monitored before every treatment cycle, during, and after treatment. Bevacizumab was discontinued if the following criteria was met: grade 4 hypertension, reversible posterior leukoencephalopathy syndrome or hypertensive encephalopathy, grade 4 nephritic syndrome, arterial thrombosis, symptomatic grade 4 or recurrent/worsening venous thromboembolic events after resumption of bevacizumab treatment, grade 3 hemorrhage, bowel perforation or fistula and any complete wound disruption.
Time Frame: 58 months
Measure: Number; unit: participants
Arm/Group | Maintenance Therapy With Bevacizumab
Number analyzed (Participants) | 15
participants
  Bowel Perforation | 1
  Leukopenia (AE grade 1-5) | 13
  Neutropenia (AE Grade 1-5) | 12
  Thrombocytopenia (AE Grade 1-5) | 9
  Anemia (AE Grade 1-5) | 15
  Allergy/Immunology (AE Grades 1-5) | 2
  Alopecia (AE Grades 1-5) | 10
  Anorexia (AE Grades 1-5) | 8
  Cough (AE Grades 1-5) | 4
  Depression (AE Grades 1-5) | 2
  Diarrhea (AE Grades 1-5) | 5
  Dyspnea (AE Grades 1-5) | 3
  Epistaxis (AE Grades 1-5) | 1
  Fatigue (AE Grades 1-5) | 12
  Gastrointestinal (AE Grades 1-5) | 9
  Hemorrhage (AE Grades 1-5) | 1
  Hoarseness (AE Grades 1-5) | 2
  Hypercalcemia (AE Grades 1-5) | 1
  Infection (AE Grades 1-5) | 2
  Lymphatics (AE Grades 1-5) | 1
  Nausea (AE Grades 1-5) | 6
  Neurosensory (AE Grades 1-5) | 6
  Ocular/Visual (AE Grades 1-5) | 1
  Pain (AE Grades 1-5) | 5
  Rash (AE Grades 1-5) | 3
  Rhinitis (AE Grades 1-5) | 1
  Tinitus | 1
  Vomiting (AE Grades 1-5) | 3

ADVERSE EVENTS:
Time Frame: 58 months
Description: Bevacizumab was to be permanently discontinued if the following criteria were met: grade 4 hypertension, reversible posterior leukoencephalopathy syndrome or hypertensive encephalopathy, grade 4 nephritic syndrome, arterial thrombosis, symptomatic grade 4 or recurrent/worsening venous thromboembolic events after resumption of bevacizumab treatment, grade 3 hemorrhage, bowel perforation or fistula and any complete wound disruption.
Arm/Group | Maintenance Therapy With Bevacizumab
Serious Adverse Events (participants affected / at risk) | 11/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maintenance Therapy With Bevacizumab (N=15)
Neutropenia (Blood and lymphatic system disorders) | 8 (8) — AE category 4 or 5
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) — Adverse Category 4 or 5
Allergy (Immune system disorders) | 1 (1)
Gastrointestinal (Gastrointestinal disorders) | 1 (1) — Adverse events grade 4 or 5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maintenance Therapy With Bevacizumab (N=15)
Leukopenia (Blood and lymphatic system disorders) | 13 (13)
Neutropenia (Blood and lymphatic system disorders) | 4 (4) — AE category 1-3
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (8) — AE grade 1-3
Anemia (Blood and lymphatic system disorders) | 15 (15) — Grade 1-3
Allopecia (Skin and subcutaneous tissue disorders) | 10 (10) — Grade 1-3
Anorexia (Gastrointestinal disorders) | 8 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) — Grade 1-3
Depression (Psychiatric disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 5 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)

LIMITATIONS AND CAVEATS:
Accrual to the study was discontinued due to the initiation of a national randomized phase II trial which included paclitaxel, carboplatin and bevacivumab with maintanence bevacizumab as one of the study arms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No